CLINICAL TRIAL: NCT04856020
Title: Role of Gray Scale and Color Doppler Ultrasound in Diagnosis of Pediatric Neck Masses
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Monica Sobhy Khalaf Boles, Principal investigator, Assiut University
Other Study IDs: Us in pediatric neck masses
Record Dates: First submitted 2021-02-12; First posted 2021-04-22 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Pediatric Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our aim is to assess the role of the gray scale and color Doppler ultrasound in diagnosis of the different pediatric neck masses .

DETAILED DESCRIPTION:
Neck masses are a common occurrence in the pediatric population and often represent a diagnostic challenge for the clinician involved . fortunately , the vast majority of these lesions are ultimately proven to be benign in nature (1).

Even though clinical examination and patient's history are the first and indispensable steps in the initial diagnosis, the role of imaging is crucial, not only to determine whether a mass represents a true tumour or not , but also to achieve a more correct diagnosis and determine the extension of the lesion and its relation with the nearby anatomic structures (2).

Ultrasound (US) should serve as the primary initial imaging modality in children for palpable masses and assessment of superficial glandular structures. Because of the smaller neck size and less subcutaneous fat, sonographic penetration and resolution is generally improved as compared with adults (3 ).

Doppler imaging can also elucidate how flow is distributed within a mass may have diagnostic significance and help us in determining the nature of the lesion as well as it is of great importance in assessment of vascular lesions (4)

Though ultrasound is most common method used for evaluation of pediatric neck masses , and CT as well as MRI are used as an additional tool when necessary ( 3 ) , few studies have looked at the sensitivity and specificity of the different imaging modalities of the pediatric neck masses and most studies have investigated the epidemiology of the pediatric neck masses (5) which make histopathological diagnosis still the gold standard in distinguishing the etiology of pediatric neck masses and ruling out malignant disease (6)

ELIGIBILITY:
Inclusion Criteria:

- Clinical cases who are suspected for and provisionally diagnosed for "neck swelling" in children (below age of 18 years).

Exclusion Criteria:

1. Patients with conditions that may hinder ultrasound examination like subcutaneous emphysema and thick skin scarring.
2. Patients who are unwilling/uncooperative or have not given consent for participation.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pediatric patients with neck masses attending at outpatient clinics at assiut university pediatric hospital.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Using gray scale ultrasound to determine the consistency of neck masses in children. | baseline
  determination if the lesion is solid (hyperechoic, hypoechoic or isoechoic in comparison to adjacent neck muscles) or cystic (anechoic) or mixed in consistency.
determination of the extension of neck masses in children. | baseline
  through assessment of height, length and width in centimeters.
determination of the definition of neck masses in children, | baseline
  whether it is well defined (rounded, oval or lobulated) , ill-defined(speculated or irregular).
using color doppler ultrasound in assessment neck masses in children. | baseline
  increased or decreased vascularity depending on number of vessels and the nature of color wave (arterial or venous),

CONTACTS AND LOCATIONS:
Overall Officials: Samy AbdElAziz, PhD, Study Chair — Assiut University; Hazem Abo Zeid, PhD, Study Director — Assiut University

REFERENCES:
- [Background] Riva G, Sensini M, Peradotto F, Scolfaro C, Di Rosa G, Tavormina P. Pediatric neck masses: how clinical and radiological features can drive diagnosis. Eur J Pediatr. 2019 Apr;178(4):463-471. doi: 10.1007/s00431-018-3305-9. Epub 2019 Jan 14. PMID 30643937
- [Background] Toma P, Esposito F, Granata C, Paolantonio G, Terranova MC, Lo Re G, Ferrara D, Rollo M, Zeccolini M, Salerno S. Up-to-date imaging review of paediatric soft tissue vascular masses, focusing on sonography. Radiol Med. 2019 Oct;124(10):935-945. doi: 10.1007/s11547-019-01050-8. Epub 2019 Jun 11. PMID 31187354
- [Background] Friedman ER, John SD. Imaging of pediatric neck masses. Radiol Clin North Am. 2011 Jul;49(4):617-32, v. doi: 10.1016/j.rcl.2011.05.005. PMID 21807165
- [Background] Stern JS, Ginat DT, Nicholas JL, Ryan ME. Imaging of pediatric head and neck masses. Otolaryngol Clin North Am. 2015 Feb;48(1):225-46. doi: 10.1016/j.otc.2014.09.015. PMID 25439556